CLINICAL TRIAL: NCT06050499
Title: Chemical Analysis of Limb Microfluidics
Acronym: CALM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: The Drummond Foundation (RAMC charity) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20SM5770; IRAS (Other: 272853)
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Limb Ischemia; Compartment Syndrome of Leg
Keywords: Microfluidics; Compartment syndrome; Limb ischaemia
MeSH Terms: conditions — Compartment Syndromes | interventions — Biosensing Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Irreversible ischaemia: patients undergoing elective amputation of a limb (e.g. peripheral vascular disease)
  Interventions: Device: Microdialysis catheter + biosensor
- Reversible ischaemia: patients undergoing an operation with a limb tourniquet or intentional controlled reduction in blood flow to the lower limb (e.g. aortic cross clamping for vascular surgery).

INTERVENTIONS:
Device: Microdialysis catheter + biosensor — Microdialysis catheter from linton instrumetal "63 MD Catheter"
  Groups: Irreversible ischaemia

SUMMARY:
Compartment syndrome (CS) is a condition where an increase in pressure in an anatomical compartment (e.g. the lower leg) affects the blood supply of the tissues, leading to tissue damage. The condition is difficult to diagnose, and more difficult to determine when and how to manage it.

Treatment aims to reduce the pressure in the compartment by whatever means possible. Surgical management by of CS is highly invasive and has associated risks including infection, damage to local structures (i.e. nerves), and possibly the inability to close the wound leading to the need for further reconstructive procedures.

The clinical challenge in suspected CS is knowing if and when to intervene. Some cases of mild CS may resolve without an operation, and therefore intervening too soon causes unnecessary harm to the patient. However, waiting too long to operate with high compartmental pressures may lead to irreversible damage to the tissues, resulting in either a useless limb or necrotic tissue needing amputation.

Current strategies for determining limb health include interrogation of symptoms, signs on examination, and serial measurements of compartmental pressures, but no absolute measurement of tissue health. As such, there is an element of clinical judgment in management and no evidence base with which to develop clear treatment guidelines. There is a need for a minimally invasive method of continuously monitoring tissue health to improve the understanding of CS and its management before significant improvement in patient outcomes can be delivered.

It is proposed the application of leg "microfluidics" - analysis of samples of leg fluid - in a series of predictable clinical scenarios which simulate the threatened and unsalvageable limb. This is with an ultimate aim of developing a method of limb fluid sampling that can predict if CS is present and requires intervention.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (aged greater than or equal to 18 years) who are either:

i. Undergoing an intervention where there is a controlled reduction in blood flow to the limb that is reversible (e.g. using a tourniquet or clamp) or irreversible (e.g. during limb amputation).

ii. At risk of developing compartment syndrome following trauma or surgical intervention as determined by the clinical care team.

Exclusion Criteria:

Age <18 years old Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged greater than or equal to 18 years) who are either:
  i. Undergoing an intervention where there is a controlled reduction in blood flow to the limb that is reversible (e.g. using a tourniquet or clamp) or irreversible (e.g. during limb amputation).
  ii. At risk of developing compartment syndrome following trauma or surgical intervention as determined by the clinical care team.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Relative concentrations of key metabolites | 20 minutes (real time analysis that takes 20 minutes to register from point of sampling to result)
  Relative concentrations of key metabolites (glucose, potassium, lactate) in lower limb interstitial fluid, estimated against baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No